CLINICAL TRIAL: NCT01482728
Title: A Phase 0 Pharmacodynamic Study of Dasatinib in Women With Newly Diagnosed Endometrial Cancer
Brief Title: Bristol-Myers Squibb Dasatinib Src Inhibition in Endometrial Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Linda R Duska, Attending, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15809
Record Dates: First submitted 2011-11-14; First posted 2011-11-30 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dasatinib — 100 mg dasatinib, the day before surgery and the day of surgery
  Other Names: Spyricel
Drug: Dasatinib — 200 mg dasatinib the day before surgery and the day of surgery

SUMMARY:
The purpose of this study is to see if the investigators can measure inhibition of a protein, Src (named for Sarcoma), in tissue and blood in patients with a diagnosis of endometrial cancer. Dasatinib is a drug that blocks the activity of an important protein in cancer cells called Src. The investigators can measure the blocking of Src in the bloodstream. However, the investigators do not know if measures in the bloodstream reflect blockage of Src in cancer tissue. The investigators are doing this study to try and see if the investigators can match what the investigators see in cancer tissue to what the investigators see in the bloodstream. the investigators hope that in the future, the investigators can use blood to measure protein inhibition by dasatinib instead of asking patients to undergo repeat biopsies.

DETAILED DESCRIPTION:
Endometrial cancer is the most common of the gynecologic malignancies; affecting 42,160 women in the US in 2009.1 In addition it is often a hormonally driven tumor, expressing in many cases both estrogen receptor (ER) and progesterone receptor (PR). While most endometrial cancers are treated successfully with surgery, there is still a need for new agents in the treatment of advanced or recurrent disease. One potential agent is dasatinib, since its target, Src Family Kinases (SFKs), has been implicated in the genesis of the disease. Although not extensive, increasing evidence indicates a link between SFKs and endometrial cancer. In addition one study in breast cancer presented at the American Society of Clinical Oncology (ASCO) in 2009 demonstrated that patients with ER positive breast tumors have a higher response rate to dasatinib, suggesting perhaps a synergy between hormonal therapy and dasatinib. Because of its high efficacy for inhibiting SFKs and growth of the tumor vasculature, as well as a possible effects on the ER, dasatinib is an exciting new possibility for treatment of endometrial cancers.

Questions regarding the ability of dasatinib to inhibit its primary target in tumor tissue (regardless of cancer type) and the relationship between inhibition of SFKs in tissue vs. SFKs in blood cells are also unresolved, as few correlative studies have accompanied the plethora of clinical trials assessing the efficacy of the drug in patients. Furthermore, the effect of dasatinib on the stability of the estrogen receptor in those tissues expressing the receptor (uterine and breast, particularly) is also unknown. Src kinase has been shown to physically associate with the ER and to mediate some of its rapid signaling effects in the presence of estrogen.6 If this physical association also stabilizes the receptor (which is normally degraded upon estrogen stimulation), dasatinib could affect estrogen receptor signaling in an indirect manner. In the Mayer study, all 9 controlled tumors were ER/PR+, suggesting a possible relationship between ER expression and dasatinib response.33 These are questions unexplored in patients. The goals of this study, therefore, are to address these questions and to provide insights for all appropriate cancer types into the action of dasatinib on SFK alone and on the ER in patient samples exposed to the drug. Furthermore, if inhibition of SFKs in blood cells correlates with that in tissue, future studies can utilize blood samples instead of or in addition to tissue to monitor dasatinib activity, obviating the need for extra biopsies or surgical samples for such analyses. The investigators therefore propose a Phase 0 study of dasatinib in patients with endometrial cancer who are undergoing planned hysterectomy. The purpose of this trial will not be therapeutic; the endpoints will be translational as per the Phase 0 design. Due to the potential relationship with ER expression, only endometrioid tumors will be studied, as they most frequently express this receptor (as opposed to clear cell or serous histologies, which most often do not express ER and are not estrogen related).

Given the extensive safety data now available for dasatinib the investigators plan to allow dosing up to the accepted Maximum Tolerated Dose(MTD) which is being used across the dasatinib program. Based on the preliminary data from the Blackwell trial in breast cancer34, adequate inhibition of src family kinases is questionable at doses even higher than 100 mg (although this study was done at steady-state after 4 weeks of treatment); thus it is unlikely that doses less than 100 mg will have any value. The investigators therefore plan to begin at 100 mg to demonstrate safety (and perhaps measurable src inhibition) and then escalate to 200 mg (which is more likely to result in measurable levels of interest) assuming safety. If feasible the investigators would anticipate the ability to demonstrate a dose response of our assay in both tissue and blood, which also requires testing two doses.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 and older
* Newly diagnosed primary histologically documented endometrioid adenocarcinoma of the endometrium that is being treated surgically with hysterectomy and BSO
* Performance status 0-1
* Agree to pre operative biopsy
* Adequate organ function
* Ability to take oral medication
* Negative serum pregnancy test

Exclusion Criteria:

* Prior therapy with dasatinib or any other anti-src drug
* Women with positive pregnancy test
* Any concurrent chemotherapy not indicated in the study protocol or any other investigational agent(s)
* Prisoners or subjects who are involuntarily incarcerated
* Histologic subtypes of endometrial cancer other than endometrioid
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness
* History of significant bleeding disorder unrelated to cancer
* No previous history of malignancy which required radiotherapy or systemic treatment within the past 5 years
* Pleural or pericardial effusion of any grade
* Cardiac symptoms including but not limited to angina, prolonged QTc interval, significant ventricular arrhythmia

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in levels of SFK protein activity in a) endometrial tumor tissue and b) blood induced within two different doses of dasatinib treatment. | 1 year
  In this study the change in levels of SFK protein activity in both tissue and blood will represent the measured pharmacodynamic response.

SECONDARY OUTCOMES:
Changes in levels of SFK protein activity in blood correlates with changes in levels of SFK protein activity in endometrial tumor tissue induced by two different doses of dasatinib treatment. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Linda R Duska, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Shah YM, Rowan BG. The Src kinase pathway promotes tamoxifen agonist action in Ishikawa endometrial cells through phosphorylation-dependent stabilization of estrogen receptor (alpha) promoter interaction and elevated steroid receptor coactivator 1 activity. Mol Endocrinol. 2005 Mar;19(3):732-48. doi: 10.1210/me.2004-0298. Epub 2004 Nov 4. PMID 15528270
- [Background] Biscardi JS, Maa MC, Tice DA, Cox ME, Leu TH, Parsons SJ. c-Src-mediated phosphorylation of the epidermal growth factor receptor on Tyr845 and Tyr1101 is associated with modulation of receptor function. J Biol Chem. 1999 Mar 19;274(12):8335-43. doi: 10.1074/jbc.274.12.8335. PMID 10075741
- [Background] Desouki MM, Rowan BG. SRC kinase and mitogen-activated protein kinases in the progression from normal to malignant endometrium. Clin Cancer Res. 2004 Jan 15;10(2):546-55. doi: 10.1158/1078-0432.ccr-0661-03. PMID 14760076
- [Background] Feng W, Webb P, Nguyen P, Liu X, Li J, Karin M, Kushner PJ. Potentiation of estrogen receptor activation function 1 (AF-1) by Src/JNK through a serine 118-independent pathway. Mol Endocrinol. 2001 Jan;15(1):32-45. doi: 10.1210/mend.15.1.0590. PMID 11145737